CLINICAL TRIAL: NCT00165607
Title: Randomized, Open, Parallel, Active Controlled Study on Fracture Prevention in Antiosteoporosis Treatment (OF Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA001R00
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Drug: MENATETRANONE

SUMMARY:
To investigate a new incidence and preventive effect of menatetrenone on vertebral fracture in patients with osteoporosis who were randomly assigned to either treatment arm receiving daily dose of calcium supplement as a monotherapy (calcium monotherapy group) or menatetrenone plus calcium supplement as a combination therapy (menatetrenone combo therapy group) for 36 months, followed by a 12-month follow-up observation to examine the preventive effect on the fracture risk.

ELIGIBILITY:
Inclusion Criteria:

Inpatient or outpatient is not asked. If using any anti-osteoporotic agent other than calcium preparations (i.e., contraindicated for concomitant use stipulated in the protocol of this post-marketing study), such agent must be discontinued. Even after the discontinuation, calcium dosing is permitted with a condition that the subsequent use is started after a 8-week elapse from the discontinuation.

* Patients with primary osteoporosis (diagnosed according to "Diagnostic Criteria for Primary Osteoporosis issued by the Japanese Society for Bone and Mineral Research (1995)."
* Post-menopausal patients aged 50 years or older.
* Patients who agree to participate in a 4-year follow-up observation.
* Patients who provide written informed consent.

Exclusion Criteira:

* Patients on warfarin potassium (Warfarin®) therapy.
* Patients with hypercalcemia.
* Patietns with renal calculus.
* Patients with a known history of hypersensitivity to calcium or menatetrenone preparations.
* Patients with severe complication in the hepatic, renal, gastrointestinal, cardio- and cerebrovascular system.
* Patients who underwent bilateral ovariectomy.
* Patients with radiotherapy in the pelvis or para-aortic area.
* Patients with the following X-ray findings;

  1. Patients showing osteophytes connecting with adjacent vertebral osteophytes
  2. Patients showing hyperostosis of ligament around the vertebral body
  3. Patients showing inter-body fusion
  4. Patients who experienced surgical intervention(s) in the spine
  5. Patients with scoliosis which disturbs a diagnosing of vertebral fracture
* Patients who have been treated with anti-osteoporotic agents, other than calcium preparation, within 8 months prior to the study treatment (but not applied to the following; if discontinued, non-treated, or shifted to calcium monotherapy for 8 weeks or longer before starting the study treatment).
* Patients who experienced bisphosphonates in the past.
* Patients who are likely to show insufficient absorption of liposoluble agents such as biliary atresia, impaired bile secretion, etc.
* Other patients who are judged to be ineligible for study entry by the investigator or investigator.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-04; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
New incidence of vertebral fracture at 36 months. vertebral fracture is morphological transformation.

SECONDARY OUTCOMES:
New incidence of clinical fracture (upper forelimb, femur, radius, and vertebral fracture associated with severe trauma that can cause fracture in normal bones of young adults) at 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Norio Iinuma, Study Director — Post-Marketing Clinical Research Department. Clinical Research Center
Locations (1):
- Ōmura, Nagasaki, Japan